CLINICAL TRIAL: NCT06788626
Title: Glucagon-like Peptide 1 Receptor Agonist in Acute Large Vessel Occlusion Stroke After Endovascular Treatment
Acronym: GALLOP2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wei Hu (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Organization: The First Affiliated Hospital of University of Science and Technology of China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GALLOP2
Record Dates: First submitted 2025-01-14; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Neuroprotective Drugs; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide (Experimental): Participants will receive 0.5mg semaglutide injection before (Day 0) and 1 week (Day 7) after EVT. Additionally, they will receive antiplatelet drugs, anticoagulation or combinations of these treatment modality according to national and institutional guidelines.
  Interventions: Drug: Semaglutide 0.5 mg; Other: Standard medical treatment
- Standard medical management (Placebo Comparator): Standard medical management. Participants will receive EVT, antiplatelet drugs, anticoagulation or combinations of these treatment modality according to national and institutional guidelines.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Semaglutide 0.5 mg — 0.5mg semaglutide injection before and 1 week after endovascular treatment.
  Arms: semaglutide
Other: Standard medical treatment — Standard medical management

SUMMARY:
The goal of this clinical trial is to learn if semaglutide works to treat acute ischemic stroke (AIS). It will also learn about the safety of semaglutide in AIS. The main question it aims to answer is: Does semaglutide improve the 90-days functional outcome in participants with acute large vessel occlusion who receive the endovascular treatment (EVT)? Researchers will compare semaglutide injection to non-injection to see if semaglutide works to improve the functional outcome in participants with EVT.

Participants will:

* Receive 0.5mg semaglutide injection before (Day 0) and 1 week (Day 7) after EVT , or EVT alone.
* Have additional blood test before and after EVT.
* Receive neurological assessment before EVT, Day 1, Day 3, Day 5-7 after EVT or on hospital discharge (whichever earlier), Day 90±14 after EVT. Audio or video of the assessment may be recorded if possible.
* Receive brain CT + CT angiogram + CT perfusion and MRI after EVT, where the CT scan may be repetitive.

ELIGIBILITY:
Inclusion Criteria:

1. LVO stroke at terminal ICA, M1 or dominant M2 with an LKW-to-randomization ≤24 hours
2. Age ≥ 18 years old
3. National Institute of Health Stroke Scale ≥ 6 at the time of brain imaging
4. Acute LVO stroke due to thromboembolism or intracranial stenosis
5. Patients who received computer tomographic or magnetic resonance angiography
6. ASPECTS ≥ 6 for patients with LKW-to-randomization ≤6 hours
7. Salvageable ischemic penumbra demonstrated by CT perfusion or MRI for patients with LKW-to-randomization between 6 and 24 hours
8. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion Criteria:

1. Use of intravenous thrombolytic therapy (alteplase or tenecteplase)
2. Pre-stroke mRS > 2 for patients <80 years and > 1 for patients ≥ 80 years old
3. Intracranial hemorrhage or brain tumour on initial imaging (except small meningiomas)
4. Simultaneous occlusion of bilateral anterior circulation, or both anterior and posterior circulation
5. Unstable hemodynamics on presentation that require resuscitation
6. Systolic blood pressure >185mmHg or diastolic blood pressure >110mmHg that cannot be controlled by antihypertensive drugs
7. Severe comorbid illness, e.g. terminal malignancy with life expectancy <1 year
8. Pregnant or lactating female
9. Participation in another clinical trial
10. Contraindications to GLP1-RA, including history of allergy to GLP-1RA, family or personal history of multiple endocrine neoplasia, medullary thyroid or pancreatic carcinoma, or proliferative diabetic retinopathy
11. Blood glucose <2.7 or > 22.2 mmol/L; platelet count <50x10^9 /L; INR >1.7
12. Patients with known estimated glomerular filtration rate of <30ml/min/1.73m2 or creatinine >3mg/dL (265.2µmol/L); chronic liver disease with Child's Pugh score C or above; or recurrent unexplained hypoglycemia.
13. Suspected or confirmed vasculitis of the central nervous system
14. Unable to complete 90-day follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The ordinal shift of modified Rankin Scale | 90±14 days after procedure
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death

SECONDARY OUTCOMES:
Proportion of patients with functional independence outcome (mRS 0-1) at day 90 | 90±14 days after procedure
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Proportion of patients with functional independence outcome (mRS 0-2) at day 90 | 90±14 days after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Proportion of patients with ambulatory and self-care capable outcome (mRS 0-3) at day 90 | 90±14 days after procedure
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Neurological Function of Participants Assessed by National Institute of Health Stroke Scale | Day 1, Day 3, Day 5-7 after EVT (or at discharge, when the patient is discharged on day 5-7)
  Zero indicates no stroke symptoms, 1-4 , 5-15, 16-20, 21-42 indicate minor, moderate, moderate to severe, and severe stroke, respectively.
Health-related Quality of Life of Participants Assessed by EuroQol-5 Dimension-5 Level | 90±14 days after endovascular treatment
  Participants rated themselves on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension was distributed from "no problems at all" to "very serious problems".
Activities of Daily Living of Participants Assessed by Bathel Index | 90±14 days after procedure
  10 rating items, each of which is categorized into 2-3 out of 5 levels: Unable, Needs major help, Needs help, Needs minor help, and Independent, and each item has a different score for each level. Independence was positively correlated with the final score.

OTHER OUTCOMES:
Intracranial Hemorrhage (ICH) | 48-72 hours after EVT
  ICH means Heidelberg classification 2 or above intracerebral hemorrhage with increment of NIHSS ≥ 4.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No